CLINICAL TRIAL: NCT01355458
Title: A Multicenter, Randomized Double-Blind, Vehicle-Controlled, Parallel Group Study to Demonstrate the Efficacy and Safety of CD07805/47 Gel Applied Topically Once Daily in Subjects With Moderate to Severe Facial Erythema Associated With Rosacea
Brief Title: Phase 3 Efficacy and Safety Study of CD07805/47 Topical Gel in Subjects With Facial Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.18140
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2013-09

CONDITIONS: Rosacea
Keywords: rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD07805/47 gel (Experimental)
  Interventions: Drug: CD07805/47 gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD07805/47 gel — applied topically once daily
  Arms: CD07805/47 gel
Drug: Placebo — applied topically once daily
  Arms: Placebo

SUMMARY:
Phase 3 efficacy and safety study of CD07805/47 topical gel in subjects with facial erythema associated with rosacea. The study hypothesis is that CD07805/47 gel, applied topically once daily is more efficacious than vehicle and provides an acceptable safety profile in the treatment of facial erythema associated with rosacea.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female who is at least 18 years of age or older.
2. A clinical diagnosis of facial rosacea.
3. A Clinician Erythema Assessment (CEA) score of greater than or equal to 3 at Screening and at Baseline/Day 1 (prior to the study drug application).
4. A Patient Self Assessment (PSA) score of greater than or equal to 3 at Screening and at Baseline/Day 1 (prior to the study drug application).

Key Exclusion Criteria:

1. Particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
2. Presence of three (3) or more facial inflammatory lesions of rosacea.
3. Current treatment with monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alpha agonists.
4. Less than 3 months stable dose treatment with tricyclic antidepressants, cardiac glycosides, beta blockers or other antihypertensive agents.
5. Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Chair — Galderma R&D; William Abramovits, MD, Principal Investigator — Dermatology Treatment & Research Center; Robert Bissonette, MD, Principal Investigator — Innovaderm Research Inc.; Zoe Draelos, MD, Principal Investigator — Dermatology Consulting Services, High Point NC; Kimberly Grande, MD, Principal Investigator — The Skin Wellness Center; Michael Jarratt, MD, Principal Investigator — Derm Research, PLLC; Charles Lynde, MD, Principal Investigator — Lynderm Research Inc; Robert Matheson, MD, Principal Investigator — Oregon Medical Research Center; Kappa Meadows, MD, Principal Investigator — The Education & Research Foundation, Inc.; Angela Moore, MD, Principal Investigator — Arlington Center for Dermatology; David Nieves, MD, Principal Investigator — Windsor Dermatology; Andrew Pollack, MD, Principal Investigator — Philadelphia Institute of Dermatology; Howard Sofen, MD, Principal Investigator — Dermatology Research Associates; Martin Steinhoff, MD, Principal Investigator — University of California, San Francisco; Daniel Stewart, DO, Principal Investigator — Michigan Center for Skin Care Research; Jerry Tan, MD, Principal Investigator — Windsor Clinical Research Inc.
Locations (15):
- United States (12):
  - Dermatology Research Associates, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Windsor Dermatology, East Windsor, New Jersey
  - Dermatology Consulting Services, High Point, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - The Skin Wellness Center, Knoxville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - DermResearch, Inc., Austin, Texas
  - Dermatology Treatment & Research Center, Dallas, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
- Canada (3):
  - Lynderm Research Inc, Markham, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research, Inc, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CD07805/47 Gel | Placebo
Started | 129 | 131
Completed | 127 | 127
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD07805/47 Gel | Placebo | Total
Number analyzed (Participants) | 129 | 131 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 117 | 234
  >=65 years | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.76) | 48.1 (12.81) | 48.8 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 102 | 206
  Male | 25 | 29 | 54
Region of Enrollment [Number; unit: participants]
  United States | 115 | 116 | 231
  Canada | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Composite Success
Description: Composite Success is defined as 2-grade improvement on both Clinician Erythema Assessment (CEA) and Patient Self Assessment(PSA).
Time Frame: Day 29
Population: Intent-to-Treat (ITT) population (i.e. Hours 3,6,9,12)
Measure: Number; unit: participants
Arm/Group | CD07805/47 Gel | Placebo
Number analyzed (Participants) | 127 | 128
participants
  Day 29 / Hour 3 | 40 | 14
  Day 29 / Hour 6 | 39 | 12
  Day 29 / Hour 9 | 33 | 13
  Day 29 / Hour 12 | 29 | 11
Statistical Analysis 1: Comparison: CD07805/47 Gel vs Placebo; Test type: Superiority or Other; p < 0.001, GEE: Logit link function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model

ADVERSE EVENTS:
Arm/Group | CD07805/47 Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 1/129 | 0/131
Other Adverse Events (participants affected / at risk) | 0/129 | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD07805/47 Gel (N=129) | Placebo (N=131)
Accidental drug intake by child (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Study product was accidentally ingested by two young children of a single study subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days